CLINICAL TRIAL: NCT05740930
Title: Effectiveness and Safety of Partition Multi-point Defocused Myopia Management Spectacle Lens in Myopia Control Compared With Spectacle Lenses With Aspherical Lenslets: a Randomised Non-inferiority Trial
Brief Title: Effectiveness and Safety of Partition Multi-point Defocused Myopia Management Spectacle Lens in Myopia Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023KYPJ004
Record Dates: First submitted 2023-02-08; First posted 2023-02-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Myopia
Keywords: Partition multi-point defocused; Myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants wear the partition defocus myopia management spectacle lens.
  Interventions: Other: Partition defocus myopia management spectacle lens
- Control group (Active Comparator): spectacle lenses with aspherical lenslets
  Interventions: Other: Spectacle lenses with aspherical lenslets

INTERVENTIONS:
Other: Partition defocus myopia management spectacle lens — Participants in the intervention group will receive the partition defocus myopia management spectacles lens and receive follow-up checks.
  Arms: Intervention group
Other: Spectacle lenses with aspherical lenslets — Participants in the control group will receive the spectacle lenses with aspherical lenslets and receive follow-up checks.
  Arms: Control group

SUMMARY:
Myopia is considered to be the most common type of refractive error, and the incidence of myopia has shown a trend of low age. Recent studies found that the new aspheric microlens spectacle lens can more effectively control the progress of diopter than the single-vision spectcale lens. A new technology of equivalent defocusing around the lens called the partition multi-point defocus optical technology is adopted in this study.

DETAILED DESCRIPTION:
Myopia is considered to be the most common type of refractive error, and it has increased rapidly worldwide. The vision damage caused by uncorrected myopia seriously affects the quality of life, may lead to poor academic performance of children, and cause considerable economic burden. About 90% of vision damage caused by myopia can be prevented by cost-effective interventions or treatment.

In recent years, the incidence of myopia has shown a trend of low age. Therefore, clinical intervention should be carried out in the childhood stage, which is the key period of eye development, to control the progress of myopia. A recent 2-year randomized controlled study in China found that the new aspheric microlens myopia control spectacle lens can more effectively control the progress of diopter than the single-vision spectcale lens. Different studies have found or proved the technical principle of the new aspheric defocusing microlens.

Animal experiments found that the direction, intensity and regional distribution of optical defocus signals have a substantial impact on the growth of eyes; The diopter of peripheral relative hyperopia can affect the central myopia; The changes of myopia and optical defocus in the nasal and temporal regions can change the shape and peripheral refraction of the eyes; Local changes in the effective focus of the eye will lead to regional changes in eye growth and refractive error. Based on the findings of animal experiments, the new technology of equivalent defocusing around the lens called the partition multi-point defocus optical technology is adopted in this study.

A prospective, single-center, open-label, non-inferiority randomized controlled trial is developed to evaluate the effectiveness and safety of partition multi-point defocused myopia management spectacle lens among children in China in myopia control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8 to 13 years;
* Under the condition of bilateral cycloplegic autorefraction, the spherical refractive error of -0.75 to -4.75 D in each eye and astigmatism of not more than 1.50 D and anisometropia of not more than 1.00 D;
* Best-corrected visual acuity of equal or better than 0.00 LogMAR (>= 1.0 as Snellen).
* The intraocular pressure of 10 to 21mmHg.
* Volunteer to participate in this clinical trial with signature of the informed consent form.

Exclusion Criteria:

* History of eye injury or intraocular surgery;
* Clinically abnormal slit-lamp findings
* Abnormal fundus examination
* Ocular disease, such as uveitis and other inflammatory diseases, glaucoma, cataract, fundus diseases, eye tumors, dominant strabismus, and any eye diseases that affect visual function;
* Systemic diseases causing low immunity (such as diabetes, Down's syndrome, rheumatoid arthritis, psychotic patients or other diseases that researchers think are not suitable for wearing glasses);
* Participation of the drug clinical trial within three month and the device clinical trial within one month;
* Only one eye meets the inclusion criteria;
* Unable to have regular follow-up
* Participation of any myopia control clinical research trial within three months, and currently using rigid contact lenses (including nursing products), multifocal contact lenses, progressive multifocal lenses and other specially designed myopia control lenses, atropine drugs, etc.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of spherical equivalent refraction (SER) at two years | 2 years
  The difference of SER (Diopter) at two years from baseline. SER will be measured every year after cycloplegia.

SECONDARY OUTCOMES:
Changes of axial length (AL) at two years | 2 years
  The difference of AL (mm) at two years from baseline. AL will be measured every half year by IOLMaster700.
Change of anterior chamber depth (ACD) at two years | 2 years
  The difference of ACD（mm） at two years from baseline. ACD will be measured every half year by IOLMaster700.
Change of lens thickness (LT) at two years | 2 years
  The difference of LT (mm) at two years from baseline. LT will be measured every half year by IOLMaster700.
Change of corneal power (CP) at two years | 2 years
  The difference of CP (Diopter) at two years from baseline. CP will be measured every half year by IOLMaster700.
Best corrected visual acuity at two years | 2 years
  Best corrected visual acuity measured every year by EDTRS visual acuity chart after cycloplegia.
Binocular visual function at two years | 2 years
  Binocular visual function which will be measured every year is a qualitative outcome assessed by a series of tests.
Choroidal thickness at two years | 2 years
  The difference of Choroidal thickness (μm) at two years from baseline. Choroidal thickness will be measured every year by OCTA.
Visual scale score at six months | 6 months
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2) and scaled from 0 (poor quality of life) to 100 (good quality of life).
Visual scale score at two years | 2 years
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2) and scaled from 0 (poor quality of life) to 100 (good quality of life).
Time length of wearing spectcales at two years | 2 years
  Time length of wearing spectcales collected every half year. Participants report the approximate time of wearing glasses per day and the days of wearing glasses per week.
Safty of wearing the spectacle lens | 2 years
  Safty of wearing the spectacle lens which is a qualitative outcome will be evaluated every half year by prespecified measures and definations based on symptoms and signs, intraocular pressure，slit lamp and ocular fundus checks.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfa Zeng, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Fricke TR, Holden BA, Wilson DA, Schlenther G, Naidoo KS, Resnikoff S, Frick KD. Global cost of correcting vision impairment from uncorrected refractive error. Bull World Health Organ. 2012 Oct 1;90(10):728-38. doi: 10.2471/BLT.12.104034. Epub 2012 Jul 12. PMID 23109740
- [Background] Modjtahedi BS, Abbott RL, Fong DS, Lum F, Tan D; Task Force on Myopia. Reducing the Global Burden of Myopia by Delaying the Onset of Myopia and Reducing Myopic Progression in Children: The Academy's Task Force on Myopia. Ophthalmology. 2021 Jun;128(6):816-826. doi: 10.1016/j.ophtha.2020.10.040. Epub 2020 Dec 30. PMID 33388160
- [Background] Rose K, Harper R, Tromans C, Waterman C, Goldberg D, Haggerty C, Tullo A. Quality of life in myopia. Br J Ophthalmol. 2000 Sep;84(9):1031-4. doi: 10.1136/bjo.84.9.1031. PMID 10966960
- [Background] Naidoo KS, Fricke TR, Frick KD, Jong M, Naduvilath TJ, Resnikoff S, Sankaridurg P. Potential Lost Productivity Resulting from the Global Burden of Myopia: Systematic Review, Meta-analysis, and Modeling. Ophthalmology. 2019 Mar;126(3):338-346. doi: 10.1016/j.ophtha.2018.10.029. Epub 2018 Oct 17. PMID 30342076
- [Background] Burton MJ, Ramke J, Marques AP, Bourne RRA, Congdon N, Jones I, Ah Tong BAM, Arunga S, Bachani D, Bascaran C, Bastawrous A, Blanchet K, Braithwaite T, Buchan JC, Cairns J, Cama A, Chagunda M, Chuluunkhuu C, Cooper A, Crofts-Lawrence J, Dean WH, Denniston AK, Ehrlich JR, Emerson PM, Evans JR, Frick KD, Friedman DS, Furtado JM, Gichangi MM, Gichuhi S, Gilbert SS, Gurung R, Habtamu E, Holland P, Jonas JB, Keane PA, Keay L, Khanna RC, Khaw PT, Kuper H, Kyari F, Lansingh VC, Mactaggart I, Mafwiri MM, Mathenge W, McCormick I, Morjaria P, Mowatt L, Muirhead D, Murthy GVS, Mwangi N, Patel DB, Peto T, Qureshi BM, Salomao SR, Sarah V, Shilio BR, Solomon AW, Swenor BK, Taylor HR, Wang N, Webson A, West SK, Wong TY, Wormald R, Yasmin S, Yusufu M, Silva JC, Resnikoff S, Ravilla T, Gilbert CE, Foster A, Faal HB. The Lancet Global Health Commission on Global Eye Health: vision beyond 2020. Lancet Glob Health. 2021 Apr;9(4):e489-e551. doi: 10.1016/S2214-109X(20)30488-5. Epub 2021 Feb 16. No abstract available. PMID 33607016
- [Background] He M, Zheng Y, Xiang F. Prevalence of myopia in urban and rural children in mainland China. Optom Vis Sci. 2009 Jan;86(1):40-4. doi: 10.1097/OPX.0b013e3181940719. PMID 19104465
- [Background] Wildsoet CF, Chia A, Cho P, Guggenheim JA, Polling JR, Read S, Sankaridurg P, Saw SM, Trier K, Walline JJ, Wu PC, Wolffsohn JS. IMI - Interventions Myopia Institute: Interventions for Controlling Myopia Onset and Progression Report. Invest Ophthalmol Vis Sci. 2019 Feb 28;60(3):M106-M131. doi: 10.1167/iovs.18-25958. PMID 30817829
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039
- [Background] Smith EL 3rd, Hung LF. The role of optical defocus in regulating refractive development in infant monkeys. Vision Res. 1999 Apr;39(8):1415-35. doi: 10.1016/s0042-6989(98)00229-6. PMID 10343811
- [Background] Wallman J, Gottlieb MD, Rajaram V, Fugate-Wentzek LA. Local retinal regions control local eye growth and myopia. Science. 1987 Jul 3;237(4810):73-7. doi: 10.1126/science.3603011.
- [Background] Huang J, Hung LF, Smith EL 3rd. Recovery of peripheral refractive errors and ocular shape in rhesus monkeys (Macaca mulatta) with experimentally induced myopia. Vision Res. 2012 Nov 15;73:30-9. doi: 10.1016/j.visres.2012.09.002. Epub 2012 Sep 28. PMID 23026012
- [Background] Smith EL 3rd, Hung LF, Huang J, Blasdel TL, Humbird TL, Bockhorst KH. Effects of optical defocus on refractive development in monkeys: evidence for local, regionally selective mechanisms. Invest Ophthalmol Vis Sci. 2010 Aug;51(8):3864-73. doi: 10.1167/iovs.09-4969. Epub 2010 Mar 10. PMID 20220051
- [Background] Smith EL 3rd, Hung LF, Huang J, Arumugam B. Effects of local myopic defocus on refractive development in monkeys. Optom Vis Sci. 2013 Nov;90(11):1176-86. doi: 10.1097/OPX.0000000000000038. PMID 24061154